CLINICAL TRIAL: NCT01910285
Title: Comparison of Intubation Conditions After Induction With Propofol Associated With a Dose of Remifentanil or Sufentanil in Surgical Tooth Extraction.
Brief Title: Remifentanil Versus Sufentanil for Intubation Condition Without Myorelaxant
Acronym: REMIDENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12 522 03; HAO (Other: University Hospital of Toulouse)
Record Dates: First submitted 2013-07-15; First posted 2013-07-29 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Anaesthetic Induction
Keywords: Anesthetic induction; Intubation conditions; Tooth extraction; Propofol; Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanyl- sufentanil placebo (Experimental): 3 mg/kg of propofol combined with 3 µg/kg of remifentanil
  Interventions: Drug: Remifentanyl - sufentanil placebo
- Sufentanil - remifentanyl placebo (Active Comparator): 3 mg/kg of propofol combined with 0.3 mg/kg of sufentanil
  Interventions: Drug: Sufentanil - remifentanyl placebo

INTERVENTIONS:
Drug: Remifentanyl - sufentanil placebo — Induction of general anesthesia with 3 mg/kg of propofol combined with 3 µg/kg of remifentanil and 10 ml of isotonic sodium chloride for the double blind. The trachea is then intubated after waiting the time of action of each product.
  Arms: Remifentanyl- sufentanil placebo
Drug: Sufentanil - remifentanyl placebo — Induction of general anesthesia with 3 mg/kg of propofol combined with 0.3 mg/kg of sufentanil and 25 ml of isotonic sodium chloride for the double blind. The trachea is then intubated after waiting the time of action of each product.
  Arms: Sufentanil - remifentanyl placebo

SUMMARY:
The main objective is the comparison of intubation conditions after anesthetic induction bolus of propofol-sufentanil when compared to injection of propofol-remifentanil in patients undergoing surgery for tooth extraction.

Intubation without myorelaxant with propofol and sufentanil is classic but less efficient than induction with curare on achieving perfect intubation conditions. The use of a protocol without curare is sometimes justified for short gestures or when you want to avoid allergia. Remifentanil often provides excellent intubation conditions without myorelaxant. However, remifentanil was never compared to sufentanil in terms of intubating conditions without muscle relaxant.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 to 60 years
* American Society of Anesthesiology (ASA) 1 or 2
* scheduled for surgical tooth extraction under general anesthesia with intubation
* signed consent form

Exclusion Criteria:

* criterion of difficult ventilation or intubation
* chronic alcoholism or opiate use
* beta-blockers or calcium channel blockers treatment
* allergy to paracetamol or ketoprofen
* patient under protection of justice

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Scandinavian Scale of Intubation Conditions (from Viby-Mogensen). The comparison will be made on the percentage of obtaining excellent intubation conditions. | This outcome measure is assessed at day 1 during the per-anesthetic period.

SECONDARY OUTCOMES:
percentage of patient with a decrease of over 20% in Mean Arterial Pressure (MAP) or Heart Rate (HR) | This outcome measure is assessed at day 1 during the per-anesthesic period and the monitoring period in PACU.
breath - hold time - time to extubation, time to Aldrete score of 10 in PostAnesthesia Care Unit (PACU) | This outcome measure is assessed at day 1 during the per-anesthesic period and the monitoring period in PACU.
difficult intubating scale (Adnet et al. Anesthesiology. 99) | This outcome measure is assessed at day 1 during the per-anesthesic period and the monitoring period in PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Christine ROCHE-TISSOT, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Purpan, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Indications de la curarisation en anesthésie : conférence de consensus (texte court). Ann Fr Anesth Reanim 1999;19:34-7.
- [Background] Laxenaire MC, Auroy Y, Clergue F, Pequignot F, Jougla E, Lienhart A. [Organization and techniques of anesthesia]. Ann Fr Anesth Reanim. 1998;17(11):1317-23. doi: 10.1016/s0750-7658(99)80044-6. No abstract available. French. PMID 9972359
- [Background] Laxenaire MC. [Epidemiology of anesthetic anaphylactoid reactions. Fourth multicenter survey (July 1994-December 1996)]. Ann Fr Anesth Reanim. 1999 Aug;18(7):796-809. doi: 10.1016/s0750-7658(00)88460-9. French. PMID 10486634
- [Background] Combes X, Andriamifidy L, Dufresne E, Suen P, Sauvat S, Scherrer E, Feiss P, Marty J, Duvaldestin P. Comparison of two induction regimens using or not using muscle relaxant: impact on postoperative upper airway discomfort. Br J Anaesth. 2007 Aug;99(2):276-81. doi: 10.1093/bja/aem147. Epub 2007 Jun 15. PMID 17573390
- [Background] Adamus M, Koutna J, Gabrhelik T, Zapletalova J. [Tracheal intubation without muscle relaxant--the impact of different sufentanil doses on the quality of intubating conditions: a prospective study]. Cas Lek Cesk. 2008;147(2):96-101. Czech. PMID 18383960
- [Background] Hanna SF, Ahmad F, Pappas AL, Mikat-Stevens M, Jellish WS, Kleinman B, Avramov MN. The effect of propofol/remifentanil rapid-induction technique without muscle relaxants on intraocular pressure. J Clin Anesth. 2010 Sep;22(6):437-42. doi: 10.1016/j.jclinane.2009.12.004. PMID 20868965
- [Background] Alexander R, Olufolabi AJ, Booth J, El-Moalem HE, Glass PS. Dosing study of remifentanil and propofol for tracheal intubation without the use of muscle relaxants. Anaesthesia. 1999 Nov;54(11):1037-40. doi: 10.1046/j.1365-2044.1999.00904.x. PMID 10540091
- [Background] Bouvet L, Stoian A, Rimmele T, Allaouchiche B, Chassard D, Boselli E. Optimal remifentanil dosage for providing excellent intubating conditions when co-administered with a single standard dose of propofol. Anaesthesia. 2009 Jul;64(7):719-26. doi: 10.1111/j.1365-2044.2009.05916.x. PMID 19624626
- [Background] Fujii Y, Itakura M. A comparison of pretreatment with fentanyl and lidocaine preceded by venous occlusion for reducing pain on injection of propofol: a prospective, randomized, double-blind, placebo-controlled study in adult Japanese surgical patients. Clin Ther. 2009 Oct;31(10):2107-12. doi: 10.1016/j.clinthera.2009.10.012. PMID 19922881 (Retraction: PMID 29724497 Clin Ther. 2018 Apr 30;:)
- [Background] Fattorini F, Romano R, Ciccaglioni A, Pascarella MA, Rocco A, Mariani V, Pietropaoli P. Effects of remifentanil on human heart electrical system. A transesophageal pacing electrophysiological study. Minerva Anestesiol. 2003 Sep;69(9):673-7, 677-9. English, Italian. PMID 14564237
- [Background] Maruyama K, Nishikawa Y, Nakagawa H, Ariyama J, Kitamura A, Hayashida M. Can intravenous atropine prevent bradycardia and hypotension during induction of total intravenous anesthesia with propofol and remifentanil? J Anesth. 2010 Apr;24(2):293-6. doi: 10.1007/s00540-009-0860-2. Epub 2010 Jan 26. PMID 20101512
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Egan TD, Brock-Utne JG. Asystole after anesthesia induction with a fentanyl, propofol, and succinylcholine sequence. Anesth Analg. 1991 Dec;73(6):818-20. doi: 10.1213/00000539-199112000-00025. No abstract available. PMID 1952185
- [Background] Maryniak JK, Bishop VA. Sinus arrest after alfentanil. Br J Anaesth. 1987 Mar;59(3):390-1. doi: 10.1093/bja/59.3.390. No abstract available. PMID 3103664
- [Background] Starr NJ, Sethna DH, Estafanous FG. Bradycardia and asystole following the rapid administration of sufentanil with vecuronium. Anesthesiology. 1986 Apr;64(4):521-3. doi: 10.1097/00000542-198604000-00023. No abstract available. PMID 2870669
- [Background] Wang J, Winship S, Russell G. Induction of anaesthesia with sevoflurane and low-dose remifentanil: asystole following laryngoscopy. Br J Anaesth. 1998 Dec;81(6):994-5. doi: 10.1093/bja/81.6.994-a. No abstract available. PMID 10211042
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711